CLINICAL TRIAL: NCT01727622
Title: Optimized Arterial Spin Labeling MRI for Cognitive Decline
Brief Title: Arterial Spin Labeling (ASL) MRI for Cognitive Decline
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 815471; 5R01AG040271 (NIH)
Record Dates: First submitted 2012-10-22; First posted 2012-11-16 (Estimated); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Fluorodeoxyglucose F18; Spinal Puncture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — cerebrospinal fluid
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Controls: ASL-MRI and FDG-PET will be compared for ability to discriminate between Control subjects and adults with Mild Cognitive Impairment (prodromal AD). A lumbar puncture will be obtained in a proportion of the participants.
  Interventions: Drug: FDG-PET; Other: ASL-MRI; Procedure: Lumbar Puncture
- Mild Cognitive Impairment: ASL-MRI and FDG-PET will be compared for ability to discriminate between Control subjects and adults with Mild Cognitive Impairment (prodromal AD). A lumbar puncture will be obtained in a proportion of the participants.
  Interventions: Drug: FDG-PET; Other: ASL-MRI; Procedure: Lumbar Puncture

INTERVENTIONS:
Drug: FDG-PET — Diagnostic: FDG-PET imaging to examine neuronal health
  Other Names: fluorodeoxyglucose
Other: ASL-MRI — Arterial-Spin Labeled MRI to examine cerebral blood flow
  Other Names: Arterial Spin Labeling
Procedure: Lumbar Puncture — Lumbar puncture to acquire a small amount of cerebrospinal fluid for protein level analyses. Note that this will not be required in all participants.
  Other Names: Spinal Tap

SUMMARY:
The purpose of this study is to determine the value of Arterial Spin Labeling (ASL) MRI, a measure of blood flow to the brain, in Mild Cognitive Impairment (MCI) and compare it to existing measures. In particular, the investigators will compare ASL MRI to Positron Emission Tomography (PET/CT), which measures brain metabolism reflecting how well cells in a patient's brain are functioning. In addition, the investigators will assess the relationship of these measures to specific protein levels associated with Alzheimer's Disease in the patient's cerebrospinal fluid (the fluid that surrounds the brain and spinal cord) obtained by lumbar puncture. By comparing the information that is available from these procedures to the patient's performance on cognitive tests, the investigators hope to learn which procedures most accurately reflect and assist in determination of the potential causes of cognitive difficulties that arise with MCI, and thus, which are most useful in the clinical setting. In particular, PET scans have been found to be very useful in diagnosis of MCI and Alzheimer's Disease, but the investigators want to find out if they can get the same, or better, information from an ASL MRI scan, which is less expensive and easier to acquire.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 55 and 89.
* Fluent in English
* Part of the longitudinal cohort of the PMC/ADCC (must already be or agree to become a part of the Penn Memory Center cohort so baseline neuropsychological testing is available before study participation begins)
* Adequate visual and auditory acuity to allow for neuropsychological testing
* Women: post-menopausal or surgically sterile
* Willing and able to complete all required study procedures
* Completed 6 grades of education
* Geriatric Depression scale less than 6 (assessed within 3 months)

PATIENTS ONLY:

* Diagnosis of MCI
* MMSE between 24 and 30
* Has a study partner

Exclusion Criteria:

* Any contraindication to MRI (i.e. presence of pacemaker, ferrous metal in the eye, severe claustrophobia that would preclude subject from completing the MRI, etc.).
* Major depression, bipolar disorder, history of schizophrenia
* History of substance abuse or dependence within the past 2 years.
* Any medical or neurological condition that, in the opinion of the investigator, would compromise the subject's safety, successful participation in, or integrity of the study.
* Pregnancy
* Recent history of poorly controlled diabetes (e.g. multiple blood glucose reports of ≥ 180 mg/dl.)
* Currently receiving medical or drug treatment contraindicating protocol participation e.g. anticoagulants such as Coumadin/Warfarin

Ages: 55 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This project will focus on a population enriched in individuals with incipient AD (i.e. MCI). These subjects, as well as age-matched controls, will be recruited from the Alzheimer's Disease Center at the University of Pennsylania.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2012-08; Primary Completion 2018-05-11 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Composite region of interest (ROI) measure of cerebral blood flow (CBF) measured by ASL MRI versus composite ROI measure of cerebral metabolism measured by FDG PET | 2 weeks
  Our primary aim is to determine if the diagnostic accuracy of 'state-of-the art' Arterial Spin Labeling (ASL) MRI is as good as (i.e., noninferior to) the diagnostic accuracy of FDG-PET/CT in comparison of MCI patients to cognitively normal adults. To test if ASL in noninferior to FDG-PET, we will use an asymptotic z test statistic for equivalent studies described in an equation of Zhou et al. (2002). The test statistic compares the AUCs from ASL and FDG-PET/CT by appropriately accounting for the correlation between them.

SECONDARY OUTCOMES:
Prediction of longitudinal change in hippocampal volume | 1 year
  Investigators will compare ASL MRI versus FDG PET in their ability to predict disease progression based on change in hippocampal volume. Investigators will define patients as 'progressors' if they display an atrophy rate greater than one standard deviation above the mean rate for healthy controls. Investigators will again use the composite ROI for ASL sequences and FDG-PET data to determine the best single or combination of predictors of progression.
Prediction of longitudinal change in clinical status (i.e. progression to Alzheimer's Disease) | 2 years
  Investigators will compare ASL MRI versus FDG PET in their ability to predict disease progression based on conversion to clinical Alzheimer's Disease. Investigators will determine which measure best predicts conversion to clinical Alzheimer's Disease.

CONTACTS AND LOCATIONS:
Overall Officials: David A Wolk, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Memory Center, Philadelphia, Pennsylvania, United States